CLINICAL TRIAL: NCT01954823
Title: Randomized Controlled Trial for the Evaluation of the Use of an Electronic Diary by People With Multiple Sclerosis
Brief Title: Use of an Electronic Diary by People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMC-13-0065-CTIL
Record Dates: First submitted 2013-09-29; First posted 2013-10-07 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis, Patient-reported outcomes, patient diary
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- e-diary (Experimental): The study group will have assess to an e-diary developed for people with MS, through the Internet and/or smart-phones. In addition, participants will continue to receive regular care at the MS clinic
  Interventions: Device: e-diary
- no use of e-diary (No Intervention): Participants of the control group will receive regular care at the MS clinic and will and no use of the e-diary

INTERVENTIONS:
Device: e-diary — The e-diary can collect data on:
  * Medical data: information on diseases, treatments and attending physicians
  * Diary: daily report of drugs intake, symptoms and their intensity and additional relevant data
  * Reminders: the application can send reminders on drug intake or medical appointments to cellular phones or emails
  * Reports: textual and graphical reports of the data in the diary can be created
  Arms: e-diary

SUMMARY:
Multiple Sclerosis (MS) is the most common chronic neurological disease affecting young adults, with onset usually at the age 20-40. Disease modifying therapies are available to MS, as well as drugs to improve patients' symptoms.

Choosing the optimized treatment for each patient is a challenge to neurologists since predictive biomarkers for therapy are yet to be validated and approved. Current therapy decisions are based predominantly on clinical evaluation of disability and disease relapses. Adherence to treatment in MS is sub-optimal.

Over the past few years a growing involvement of patients in their healthcare is noted, specially in chronic diseases, and Patient Reported Outcomes (PRO) are being incorporated as part of therapy evaluation.

Several electronic patients diaries to track adherence to therapy, PRO and drugs side effects in diseases such as epilepsy are available. A mobile interactive patient diary (e-diary) tailored for persons with MS was developed. Users can enter data on drugs intake, drugs-side effects and disease symptoms and receive reminders regarding adherence to treatment.

The aim of this study is to assess the benefits of the use of an e-diary for MS patients on healthcare. In order to achieve this goal, 80 MS patients will be randomized into two groups: a study group with access to the e-diary and a control group. After a period of one year, satisfaction with the e-diary will be assessed. The effect of the use of the e-diary on quality of life, on clinical outcomes and on adherence to therapy will be evaluated by comparing the two groups.

This study will indicate the possible contribution of an e-diary for the evaluation of drugs safety and efficacy and of patient adherence to therapy, to be applied in clinical trials and towards improvement of MS patient' care.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is the most common chronic neurological disease affecting young adults, with onset usually at the age 20-40. Women are affected 3-4 times more than men. The disease is characterized by 2 main phenotypes: relapsing-remitting or progressive course.

MS is a complex multi-factorial disease, with underlying both genetic and environmental factors. Different populations have different susceptibility (Compston and Coles 2008).

Clinical disability is due to distraction of the Central Nervous System (CNS) myelin (mainly oligodendrocytes) due to 3 processes (Franklin 2002; Franklin and Ffrench-Constant 2008; Frischer, Bramow et al. 2009):

1. Inflammation- immune cells with aberrant activity invade the brain and spinal cord and cause distraction of CNS myelin (process called demyelination and secondary neurodegeneration - axonal and neuronal loss)
2. Primary neurodegeneration (axonal and neuronal loss) - without prominent inflammation
3. Repair - the inflammatory and neurodegenerative processes are followed by an attempt of the CNS to repair - however, this partial and incomplete repair is often the basis of residual deficits and disability (Chandran, Hunt et al. 2008) .

These processes cause damage of the CNS, brain and spinal cord, leading to deficiencies in several neurologic systems such as motoric, sensory, sphincters, visual and cognitive.

MS is diagnosed by a clinical evaluation of the neurologist in conjunction with the detection of inflammation in the white matter in the CNS through MRI.

Following the increased understanding of the disease, in the last 10-15 years there are new subcutaneous injection immunotherapies available (COPAXON / TEVA; Interferon -beta: Avonex. Betaferon and Rebif) and Tysabri infusion . These drugs can cause side effects at such an extent that treatment may have to be discontinued. Recently an oral drug Gilenya was released to the market, and additional oral drugs such as Laquinimod and BG-12 (Dimethyl Fumarate) are at different phases of development. However these can attenuate the disease (reduce the number of relapses per year) but cannot cure it. Also, they are beneficial in only ~40 % of the Relapsing -Remitting patients. Currently there are no treatments for patients with the Progressive Disease - who have gradual increased disability (Murray 2006).

Intravenous steroids are the short term treatment for acute relapses. In addition to the long term immunomodulatory drugs, disease modifying drugs (DMD), there are also drugs used to alleviate some of the MS symptoms, such as Provigil, for fatigue and Fampyra for improvement of walking disabilities.

With the growing number of drugs available for the treatment of MS and its symptoms, the evaluation of treatment success is essential so the best treatment can be fitted to each individual. Presently, there are no objective tools for assessment of treatment efficiency. MRI is an expensive procedure that does not add much information beyond the clinical exam. CSF (cervical spine fluid) is an invasive and painful examination which can help in MS diagnosis but is not related to disease course. Treatment evaluation is based mainly in two parameters: disability (measured by EDSS) and annual relapse rate. Both measures have disadvantages: 1) EDSS indicates mostly motorical disability and does not take into account other implications of the disease, such as cognitive problems and fatigue, 2) the number of relapses per year may differ among neurologists, since generally only relapses with indication to steroids treatment are taken into consideration and steroids indication variates among neurologists.

Over the past few years a growing involvement of patients in their healthcare can be noted. Healthcare organizations recognize the importance of this involvement both because of an increasing public demand and because patient involvement is being considered positive to the health system, specially in chronic diseases.

Patient Reported Outcome-PRO can be defined as "evaluation of treatment success based on the patient point of view". The patient grades the intensity of symptoms related to the disease or side effects of the treatment and report his general well being with the help of measures such as Health-Related Quality of Life (HRQoL). PRO can be an useful measure in treatment evaluation for some reasons: First, patients today expect to know about drugs side effects not only from the medical staff point of view but also from the view of other patients taking the drug (Basch 2010). Secondly, one of the bigger challenges today in the management of MS is treatment adherence. It has been shown that about 50% of the patients discontinue disease modifying therapy before completing two years of treatment (Bruce and Lynch 2011). PRO could contribute to the identification of the reasons for non-adherence allowing interventions for adherence improvement.

The main difficulties for collecting PRO are: 1) the patient capability of relating to the physician during an encounter all the relevant symptoms he had since the last visit, and 2) the fact that the patient's report has to be compared to his adherence to therapy. Recently the FDA, recognizing the importance of the use of PRO, has founded a consortium for developing and evaluating PRO (Riazi 2006; Goldman 2010).

An electronic diary (e-diary) tailored for persons with MS was developed. The diary is an Internet application that can be used through the web or iphones. Data on medical history, drugs intake, drugs side effects and disease symptoms (including intensity) can be entered by the user. The application can produce graphs based on the data entered and send reminders to the user's email or cellular phone. It can give the physician a complete insight on patient adherence and on the outcomes according to the patient's view.

A similar diary for persons with epilepsy has been used by thousands of persons in the past two years (https://my.epilepsy.com/irody/login-page.php) (Fisher 2010; Le 2011). In face of the importance of patient involvement in medical decisions and since that are not objective measures of treatment success in Multiple Sclerosis that can be used routinely, an electronic diary can contribute to the evaluation of therapy, regarding both efficiency and safety.

Aim(s)

The main aims of this study are to assess the contribution of the use of an e-diary by people with MS on:

1. Adherence to therapy;
2. Quality of life and clinical outcomes; and
3. Collection of data on disease symptoms, treatment side-effects, and PRO and its relevance for clinical decision making.

A second aim of this study is to assess the e-diary usability.

Research hypothesis Patient use of an electronic diary will contribute to patient adherence to treatment and to clinical outcomes and will allow collection of reliable data on symptoms, side effects and treatment outcome from the patient point of view.

Work plan outline:

MS Patients, visiting the Multiple Sclerosis Center at the Carmel Medical Center and being treated by DMD or symptomatic drugs for MS will be invited to participate in this study. After recruitment and signing an informed consent for the study, participants will be randomized in two groups: the first one, the study group, will have access to a MS patients e-diary during one year, and in parallel will continue to receive standard medical follow-up. The second one, the control group, will receive standard medical care only. Participants of both groups will be asked to fill questionnaires on demographic data, quality of life and therapy adherence.

The e-diary allows data entry and retrieval through computers or iPhones. Users can enter data on medications, medical visits, drugs side effects, receive reminders and produce graphic and textual reports of the data entered. Participants will use the diary for one year and details of the use will be automatically collected. In the end of this period, clinical and personal data of each group on baseline and after one year and of the two groups will be compared. Users' and medical team satisfaction of the e-diary will be evaluated.

Study plan:

Number of participants: 100 MS patients.

MS patients will be recruited through the MS center clinic at Carmel Medical Center after receiving an explanation from Prof. Miller, or the attending neurologist authorized by Prof Miller to do so, on the study aims and protocol, and signing an informed consent, including the release of Clalit Health Services from any responsibility regarding information security. Participants will be randomized in two groups: the first one, the study group, will have access to a MS patients e-diary during one year, and in parallel will continue to receive standard medical follow-up. The second one, the control group, will receive standard medical care only. Information regarding their personal and family medical history, including data such as demographic and ethnicity data, data on smoking and dietary habits, vitamins intake, other diseases, education and occupation will be collected from both groups via the "Personal information questionnaire". Participants will also fill the MSTAQ (Multiple Sclerosis Treatment Adherence Questionnaire) questionnaire on adherence to treatment at baseline, after 6 months and one year, and the MSQoL-54 (Multiple Sclerosis Quality of Life-54 Instrument) questionnaire on quality of life at baseline and after one year. Medical staff will fill the "Clinical questionnaire" detailing patient clinical status prior to the study and the Clinical Follow-up questionnaire" after 6 months and one year. These questionnaires will be filled in printed forms during participants visits to the clinic. When necessary, data will also be collected from medical records. Data collected through participants and physician filled forms and from medical records will be stored on an Excel or Access data base. In addition, data regarding the use of the diary will be automatically collected.

Use of the electronic diary:

Participants in the study group will receive a code to access the e-diary through a computer or an iPhone. Participants that don't have an I-phone may be granted one for the study period. The data entered in the diary will be maintained in a secured Internet server and will not include any identified data.

The diary can collect data on:

* Medical data: information on diseases, treatments and attending physicians
* Diary: daily report of drugs intake, symptoms and their intensity and additional relevant data
* Reminders: the application can send reminders on drug intake or medical appointments to cellular phones or emails
* Reports: textual and graphical reports of the data in the diary can be created The e-diary was developed for patient use and data entered is not automatically accessed by the medical staff. Patients will be instructed to bring the reports produced by the diary to their medical appointments. In addition, patients will be instructed to contact by phone the medical staff at the clinic in case they feel any change and/or deterioration in their medical condition, as habitual in our clinic.Participants of the study group will receive instructions on how to use the diary and technical assistance will be available during the study. Follow-up on diary's use will take 1 year. The medical follow-up of participants will be as usual in the MS center for both groups.

Data regarding the use of the diary will be collected directly from the application, including:

* Number of entries
* Duration of entries
* Frequency and pattern of use
* Pages visited
* Time elapsed between a clinical event and report to the clinical staff
* Access by computer or Iphone
* Adherence to treatment
* Clinical related data Participants showing low/no access to the application will be contacted by the medical team and will be encouraged to use the diary. These contacts will be taken into consideration during statistical analysis.

After the follow-up period participants of the study group and the medical staff will fill the "Questionnaire for Diary evaluation" regarding satisfaction from the tool. Medical staff will fill the "Clinical follow-up questionnaire" for the two groups.

Data analysis

In the end of the follow-up period, data collected directly from the application and data from the questionnaires will be analyzed as follows:

1) Adherence to treatment: In the study group, adherence to treatment will be assessed by data registered on the e-diary and by questionnaires applied on baseline, after six months and one year. In the control group, adherence to treatment will be assessed by questionnaires only. Questionnaires from the two groups will be compared. In addition, the study group questionnaire on adherence will be compared to data on adherence registered in the e-diary . 2) Health-related quality of life and clinical outcomes: Clinical data such as EDSS, number of relapses and hospitalizations will be collected by questionnaires completed by the medical team. Quality of life will be assessed by questionnaires completed by the two groups on baseline and after one year and the results will be compared. Since patients can ask to visit the clinic or to call the medical team beyond regular follow-up if they feel necessary, the number of these visits and calls in the two groups will be compared. 3) Data captured in the e-diary: Data entered by the study group in the e-diary will be compared to data entered in the Electronic Medical Record by the medical team during regular follow-up of the control group. Data from both groups will be classified according to various parameters such as: relating to efficacy or safety of therapy, physician response and physical or emotional symptom. 4) E-diary usability: Adherence to the diary will be assessed from data on the pattern of use of each participant. Satisfaction will be assessed through questionnaires applied both to patients and to attending physicians.

Ethical issue:

Treatment will not be affected by participation in the study. Data collection and handling will be coded to assure privacy of participants and will be handled by Prof. Ariel Miller and his authorized staff. All the keys to the codes will be saved. Participants' regular follow-up and visits to the clinic will continue.

Data management:

Data collected through participants and physician filled forms and from medical records will be stored in an Excel or Access data base. The database is password protected, Prof Ariel Miller, and his authorized staffs are responsible for its update and data verification.

Statistics:

The continuous variables will be presented by mean, median and standard deviation. The categorical variables will be presented in percentages. Differences in demographic and clinical characteristics between the study group and the control group will be assessed using Chi square test for the categorical variables, Independent t-test or Mann Whitney, as appropriate, for the continuous variables. Differences in each group separately between baseline and after 1 year will be assessed using McNemar test for the categorical variables, paired T-Test or Wilcoxon paired test, as appropriate, for the continuous variables. For more than two time points, Friedman test will be used. Multivariate logistic regression will be used to identify which variables are independently associated to an increase in adherence.Values p<0.05 will be considered to be significant.

Timetable:

The proposed study is scheduled for two years. Follow-up on the use of the electronic diary will take up to one year and afterwards the data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* MS patients visiting the MS clinic in the Carmel Medical Center, Haifa, Israel, that are currently receiving, or, are about to receive immunomodulatory treatment or/and receiving treatment for MS symptoms.
* Patients that browse in the Internet.
* Willing and able to give inform consent
* Age 18 to 70 years

Exclusion Criteria:

* Technical difficulties in the use of an e-diary

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Adherence to therapy | one year
  Adherence to therapy will be assessed through questionnaires on adherence in the study group and in the control group, at baseline and after one year.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Miller, MD/PhD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Le S, Shafer PO, Bartfeld E, Fisher RS. An online diary for tracking epilepsy. Epilepsy Behav. 2011 Dec;22(4):705-9. doi: 10.1016/j.yebeh.2011.08.035. Epub 2011 Oct 4. PMID 21975298
- See also: Related Info — http://humanepilepsyproject.org/